CLINICAL TRIAL: NCT01858415
Title: Evaluation of Safety and Efficacy of TriPollar Device for Treatment of Wrinkles and Rhytides
Brief Title: Evaluation of Safety and Efficacy of TriPollar Device for Treatment of Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pollogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC210118_S, rev. 01
Record Dates: First submitted 2013-04-21; First posted 2013-05-21 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Facial Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Device: TriPollar

INTERVENTIONS:
Device: TriPollar

SUMMARY:
The TriPollar is intended for non invasive treatment of facial wrinkles and rhytides. This study was designed in order to evaluate the safety and efficacy of the TriPollar.

DETAILED DESCRIPTION:
The TriPollar technology is based on three or more electrodes designed to deliver RF current focused into the skin, thus generating heat in the dermal layer. Selective and focused electro-heating of the skin is intended to stimulate collagen remodeling in the dermal layer resulting in non invasive wrinkle treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject read, discussed and signed the Consent Form,
* Healthy female/male aged 35 65 years,
* Has facial wrinkles,
* Capable of reading, understanding and following instructions of the procedure to be applied,
* Able and willing to comply with the treatment and follow-up schedule.

Exclusion Criteria:

* Listed in approved protocol, and ICF

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety of TriPollar | 6 months
  Safety will be established by physician's assessment/observation of adverse events.
Efficacy of TriPollar | 6 months
  Efficacy will be established by level of wrinkle reduction at 3 m fu based on photos evaluation by independent physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Barki, PhD, Study Director — Pollogen
Locations (2):
- United States (2):
  - Ronald L Moy, Inc., Beverly Hills, California
  - Reaserch Across America, Plano, Texas